CLINICAL TRIAL: NCT06535945
Title: Influence of Human Albumin Supplementation on Kidney Dysfunction After Liver Transplantation
Acronym: HALT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC22_9739_HALT; 2024-514804-14-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Liver Transplantation; Acute Kidney Injury
Keywords: Liver; Transplantation; Albumin; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 g/L or below (Experimental): Receive Human Albumin 20% Solution when albumin serum concentration is at 30 g/L or below
  Interventions: Drug: Albumin administration
- 20 g/L or below (Active Comparator): receive Human Albumin 20% Solution when albumin serum concentration is at 20 g/L or below
  Interventions: Drug: Albumin administration

INTERVENTIONS:
Drug: Albumin administration — when albumin serum concentration is at 30 g/L or below

SUMMARY:
To verify whether albumin administration to achieve serum concentration above 30g/L (treated group) and its maintenance within plasmatic physiologic range (above 30 g/L) for five days diminishes rate of AKI at Day 7 after liver transplantation as compared to restrained albumin administration (when serum concentration is at 20 g/L or below (control)).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects equal or above 18 yrs old.
* Recipients of primary liver allografts from a deceased donor (including after cardiac death) and as a single organ (liver only).
* Capability of understanding the purpose and risks of the study.
* Written informed consent

Exclusion Criteria:

* Fulminant hepatitis
* Kidney injury at baseline (Estimated Glomerular Filtration Rate < 50 ml/min in Modification of diet in renal disease-6) including hepatorenal syndrome
* Use of an induction agent Basiliximab at liver transplantation
* Protected person (adults legally protected, under judicial protection, guardianship, or supervision), person deprived of their liberty
* At the time of randomisation, participation to another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2028-04-26 (Estimated); Study Completion 2028-04-26 (Estimated)

PRIMARY OUTCOMES:
Acute Kindey Injury at Day 7 | 7 days after liver transplantation
  To verify whether albumin administration to achieve serum concentration above 30g/L (treated group) and its maintenance within plasmatic physiologic range (=30 g/L) for five days diminishes rate of Acute Kindey Injury at Day 7 after liver transplantation as compared to restrained albumin administration (when serum concentration is at 20 g/L or below (control)).

SECONDARY OUTCOMES:
Occurrence and Severity of each Acute Kindey Injury during the first 7 days after liver transplantation | 7 days after liver transplantation
  Occurrence and Severity of each Acute Kindey Injury during the first 7 days after liver transplantation
hospital length of stay | 28 days
  hospital length of stay
occurrence of calcineurin inhibitor induced neurotoxicity | 28 days
  occurrence of calcineurin inhibitor induced neurotoxicity
occurence of calcineurin inhibitor withdraw | 28 days
  occurence of calcineurin inhibitor withdraw
occurrence of postoperative infections | 28 days
  occurrence of postoperative infections
occurrence of acute graft rejection | 28 days
  occurrence of acute graft rejection
occurrence of early graft dysfunction | 28 days
  occurrence of early graft dysfunction
duration of mechanical ventilation | 28 days
  duration of mechanical ventilation
reintubation rate | 28 days
  reintubation rate
Intensive Care Unit length of stay | 28 days
  Intensive Care Unit length of stay
Intensive Care Unit readmission rate | 28 days
  Intensive Care Unit readmission rate
All cause mortality | 28 days
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Pauline HOUSSEL-DEBRY, MD, Principal Investigator — CHU Rennes
Locations (8):
- France (8):
  - 08_CHRU de Tours Hôpital Trousseau, Chambray-lès-Tours
  - 03_APHP Hôpital Beaujon, Clichy
  - 04_CHU de Lille Hôpital Huriez, Lille
  - 05_HCL Hôpital de la Croix Rousse, Lyon
  - 06_CHU de Montpellier Hôpital St Eloi, Montpellier
  - 02_CHU de Bordeaux - Hôpital Haut Leveque, Pessac
  - 01_CHU de Rennes Hôpital Pontchaillou, Rennes
  - 09_APHP Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: European Medicines Agency Registry — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2024-514804-14-00